CLINICAL TRIAL: NCT04012333
Title: The Effect of Higher Protein Dosing in Critically Ill Patients: A Multicenter Randomized Trial
Acronym: EFFORTcombo
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: PI left site
Sponsor: RWTH Aachen University (Other)
Collaborators: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18-108
Record Dates: First submitted 2019-07-03; First posted 2019-07-09 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Nutritional Disorder; Critical Illness; Malnutrition; Frailty; Sarcopenia
MeSH Terms: conditions — Nutrition Disorders; Critical Illness; Malnutrition; Frailty; Sarcopenia

STUDY DESIGN:
Intervention Model Description: Intervention: enteral and parenteral nutrition to reach protein target of 2.2g/kg/day Control: only enteral nutrition to stay below protein target of 1.2g/kg/day
Who Masked: Outcomes Assessor
Masking Description: Study staff performing the functional outcome measurements will be blinded to study treatment group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients will receive standard care plus OLIMEL 7,6%E or if no central venous access available PeriOLIMEL 2,5%E to reach protein targets: >2.2g/kg/day
  Interventions: Drug: OLIMEL 7,6%E / PeriOLIMEL 2,5%E
- Standard Care (No Intervention): Patients will receive standard care (enteral nutrition only) to stay below the protein level: <1.2g/kg/day

INTERVENTIONS:
Drug: OLIMEL 7,6%E / PeriOLIMEL 2,5%E — OLIMEL 7,6%E will be administered via a central access whereas PeriOLIMEL 2,5%E will be administered peripherally.
  Arms: Intervention

SUMMARY:
The primary research question: In critically ill patients with nutrition 'risk factors', what is the effect of providing combined EN/PN to the group prescribed a higher dose (≥2.2 grams/kg/day) of protein/amino acid administration compared to a low group prescribed ≤1.2 gram/kg/day (EN only) on patient's functional recovery as measured by 6-minute walk distance just prior to hospital discharge? The hypothesis: Compared to a control group reflective of usual care prescribing practices and an EN only approach, the administration of a higher dose protein/amino acids using EN and PN to nutritionally high-risk critically ill patients will be associated with improved functional outcome.

DETAILED DESCRIPTION:
Positive, neutral, or negative, the results of the EFFORTcombo study will inform the clinical practice in ICU settings around the world. If positive, because of the pragmatic, multicentre nature of this trial, results will be broadly applicable to all critically ill patients worldwide. If the results are negative, it will be ensured that patients no longer receive high-dose protein/amino acid admixtures or possibly, combined EN/PN.

As it relates to critical care nutrition practice in general, there is a long history of practice-changing initiatives. A process of synthesizing (in the form of evidence-based clinical practice guidelines) and disseminating best practice ideas (in the form of web-based repository of tools and information [see www.criticalcarenutrition.com]) was established.

Over the past several years, this program of research with leaders of the American Society of Parenteral and Enteral Nutrition (ASPEN) and this specific protocol at the annual Clinical Nutrition Week with society leaders, researchers, and the clinical nutrition community at large has been discussed. Partnership with ASPEN will further facilitate both, recruitment initiatives and, importantly, the knowledge translation initiatives. These efforts will increase the likelihood of the uptake of EFFORT results across the world.

This study has both the potential to answer a high-priority clinical question and also transform the new approach in clinical nutrition research. It further represents a unique collaboration between ASPEN, its global partners, and the Clinical Evaluation Research Unit, a methodological support center based in Kingston, Ontario, Canada and managed by Dr. Daren Heyland. If successful, this type of collaboration sets an important precedent for how this community may approach additional research questions related to clinical nutrition. Nested within this larger volunteer-driven registry trial, the aim is to complete a significant sub-study that will establish the role of combined EN/PN in these nutritionally high-risk patients. This protocol pertains to the specifics of this sub-study of combined EN/PN. At the end of the trial, the data from this sub-study will be merged into the results of the overall parent EFFORT Trial (where data points are similar).

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old;
2. Expected to remain mechanically ventilated for an additional 48 hours from screening;
3. And have one or more of the following risk factors that make them at high nutritional risk:

   1. Low (≤25) or High BMI (≥35)
   2. Moderate to severe malnutrition (as defined by local assessments). We will document the means by which sites are making this determination and capture the elements of the assessment (history of weight loss, history of reduced oral intake, etc.).
   3. Frailty (Clinical Frailty Scale 5 or more from proxy)
   4. Sarcopenia (SARC-F score of 4 or more from proxy)
   5. From point of screening, projected duration of mechanical ventilation >4 days

Exclusion Criteria:

1. >96 continuous hours of mechanical ventilation before enrollment
2. Expected death or withdrawal of life-sustaining treatments within 7 days from screening
3. Pregnancy
4. The responsible clinician feels that the patient either needs low or high protein
5. Absolute contraindication to EN
6. Severe metabolic disorders including electrolyte disorders, uncontrolled hyperglycemia, hyperlipidemia, hypophosphatemia.
7. Severe chronic liver disease (MELD-score >20) or acute fulminant hepatitis.
8. Metabolic disorders involving impaired nitrogen utilization
9. Not ambulating independently prior to illness that lead to ICU admission (use of gait aid permitted)
10. Lower extremity injury or impairments that prevents them walking prior to hospital discharge (e.g. amputation, knee/hip injury)
11. Pre-existing cognitive impairment or language barrier that prohibits outcomes assessment
12. Pre-existing primary severe systemic neuromuscular disease resulting in severe weakness pre-ICU (e.g., Guillain Barre)
13. Intracranial or spinal process affecting motor function
14. Patients in hospital >5 days prior to ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
6-minute walking distance | at hospital discharge, up to 12 weeks
  measured by performing a 6-minute walking test

SECONDARY OUTCOMES:
Overall strength-upper and lower extremity | at hospital discharge, up to 12 weeks
  MRC sum-score
Quadriceps force-lower extremity strength | ICU and at hospital discharge, up to 12 weeks
  Hand held dynamometry
Distal strength-hand grip strength | ICU and at hospital discharge, up to 12 weeks
  Hand grip dynamometry
Overall Physical Functional status | Baseline (questionnaire only) and SPPB & FSS- ICU at ICU and at hospital discharge, up to 12 weeks
  Walking Impairment Questionnaire
Overall Physical Functional status | Baseline (questionnaire only) and SPPB & FSS- ICU at ICU and at hospital discharge, up to 12 weeks
  FSS-ICU
Overall Physical Functional status | Baseline (questionnaire only) and SPPB & FSS- ICU at ICU and at hospital discharge, up to 12 weeks
  SPPB
Discharge location | at hospital discharge, up to 12 weeks
  Discharge location
Body composition | Enrollment, ICU day 10 and at hospital discharge, up to 12 weeks
  Ultrasound of quadriceps
Body composition (when clinically available) | Only when clinically available, from 2 weeks before enrolment until 2 weeks after enrolment
  Abdominal CT scan at 3rd lumbar vertebra
Health-related quality of life | (Telephone) survey at baseline and 6 months
  SF-36
Physical functioning | (Telephone) survey at hospital discharge, up to 12 weeks and 6 months
  Katz ADL
Health-related quality of life | (Telephone) survey at 6 months
  EQ-5D-5L
Physical functioning | (Telephone) survey at 6 months
  Lawton IADL

CONTACTS AND LOCATIONS:
Overall Officials: Christian Stoppe, MD, Principal Investigator — University Hospital, Aachen
Locations (1):
- University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hill A, Heyland DK, Elke G, Schaller SJ, Stocker R, Haberthur C, von Loeffelholz C, Suchner U, Puthucheary ZA, Bear DE, Ney J, Clasen KC, Meybohm P, Lindau S, Laurentius T, Stoppe C. Meeting nutritional targets of critically ill patients by combined enteral and parenteral nutrition: review and rationale for the EFFORTcombo trial. Nutr Res Rev. 2020 Dec;33(2):312-320. doi: 10.1017/S0954422420000165. Epub 2020 Jul 16. PMID 32669140